CLINICAL TRIAL: NCT02307214
Title: Tako-Tsubo Cardiomyopathy and Cardiac Syndrome X: New Insights Into the Pathophysiology of Two Orphan Cardiac Diseases
Brief Title: Tako-Tsubo Cardiomyopathy and Cardiac Syndrome X: New Insights Into the Pathophysiology
Acronym: ENDAUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Giovanni Bellinzona (Other)
Responsible Party: Principal Investigator, Professor Augusto Gallino, Professor MD, Ospedale San Giovanni Bellinzona
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CE 2688
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Syndrome X; Takotsubo Cardiomyopathy
MeSH Terms: conditions — Microvascular Angina; Takotsubo Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Coronary X syndrome (Other): BaroReflex Sensitivity, endothelial function measurement
  Interventions: Other: BaroReflex Sensitivity, endothelial function measurement
- Tako-tsubo cardiomyopathy (Other): BaroReflex Sensitivity, endothelial function measurement
  Interventions: Other: BaroReflex Sensitivity, endothelial function measurement
- Healty Volunteers (Other): BaroReflex Sensitivity, endothelial function measurement
  Interventions: Other: BaroReflex Sensitivity, endothelial function measurement

INTERVENTIONS:
Other: BaroReflex Sensitivity, endothelial function measurement — no other
  Other Names: BaroReflex Sensitivity measurement by volume-clamp method (Finapress); Endothelial function measured by Endopat

SUMMARY:
Tako-Tsubo Cardiomyopathy (TTC) and Cardiac Syndrome X (CSX) are respectively acute and chronic cardiac conditions whose clinical presentation, mimicking the onset of acute myocardial ischemia in absence of epicardial coronary disease, has progressively gained the interest of the scientific community. However, despite significant progress, their underlying pathophysiology, which seems to evoke some similarities, still remains elusive. Endothelial dysfunction and autonomic imbalance have both been individually implied in their puzzling pathogenesis.

The investigators plan to conduct our study in a cohort of TTC patients, CSX patients and healthy volunteers with the following primary objective: to assess the response of endothelial function (through the Endopat score) to the autonomic tone activation induced by a 10-minute stress mental test. The assessment of autonomic tone during activation through the evaluation of Spontaneous BaRoreflex Sensitivity (BRS) and its correlation with endothelial function (Endopat score) will represent secondary objectives.

Our study will enroll 15 patients with TTC at least six months after the event, 15 patients with classic CSX and 15 healthy volunteers who will serve as control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the Mayo Clinic's criteria established diagnosis of TTC at least 6 month after the acute event
* Patients with CSX defined by the presence of anginal pain, positive exercise stress testing and negative coronary angiography.
* A comparable cohort of healthy volunteers age and sex-matched with patients

Exclusion Criteria:

* Short-term life-threatening pathology (life expectancy < 6 months)
* Physically unable to participate in the study
* Compliance not guaranteed
* Pregnancy
* Conditions that make BRS and Endopat measurements impossible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Difference in endothelial function in response to autonomic tone (Endopat score) | Baseline
  Difference in endothelial function assessed by Endopat score in response to autonomic tone induced by 10-minute mental stress test between the three groups (CSX, TTC, healty volunteers)

SECONDARY OUTCOMES:
BaroReflex Sensitivity (Sensitivity measurement by volume-clamp method (Finapress) | Baseline
  Changes in BaroReflex Sensitivity from baseline in three three groups (CSX, TTC, healty volunteers)
BaroReflex Sensitivity and endothelial dysfunction ( | Baseline
  Correlation with between BaroReflex Sensitivity [volume clamp method] and EndoPAT score in the three groups (CSX, TTC, healty volunteers)
Endothelial dysfunction (Changes in Endopat score) | Baseline
  Changes in Endopat score from baseline in three three groups (CSX, TTC, healty volunteers)

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Gallino, Prof MD, Principal Investigator — Ospedale Regionale di Bellinzona e Valli - Ospedale San Giovanni, Bellinzona; Mattia Cattaneo, MD, Study Chair — Ospedale Regionale di Bellinzona e Valli - Ospedale San Giovanni, Bellinzona; Alessandra Pia Porretta, MD, Study Chair — Ospedale Regionale di Bellinzona e Valli - Ospedale San Giovanni, Bellinzona
Locations (1):
- Ospedale Regionale di Bellinzona e Valli - Ospedale San Giovanni, Bellinzona, Bellinzona, Canton Ticino, Switzerland